CLINICAL TRIAL: NCT00266136
Title: Risk-stratified Therapy for Primary and Secondary AML and MDS. A Randomized Study by AMLCG in Relation to Cytogenetically Defined Prognostic Factors (1) on the Role of High-dose AraC as Part of Double Induction, (2) on G-CSF Priming, and (3) on High-dose Chemotherapy With Stem Cell Transplantation
Brief Title: Biology and Treatment Strategy of AML in Its Subgroups: Multicenter Randomized Trial by the German Acute Myeloid Leukemia Cooperative Group (AMLCG)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Büchner, Prof. Dr. Thomas Büchner MD PhD, University Hospital Muenster, University Hospital Muenster
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AMLCG 99; BMBF 01 GI 02070
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML treatment, de-novo, secondary, high-risk MDS, chemotherapy, autologous SCT, adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm Metastasis | interventions — Cytarabine; Thioguanine; Daunorubicin; Cyclophosphamide; Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Cytarabine — see protocol
Drug: Thioguanine — see protocol
Drug: Daunorubicin — see protocol
Drug: Cyclophosphamide — see protocol
Drug: G-CSF — see protocol
Procedure: Autologous stem cell transplantation — for details see protocol
Procedure: Allogeneic stem cell transplantation — for details see protocol

SUMMARY:
The study in patients with primary and secondary AML and high-risk MDS uses a risk-stratified, randomized design to evaluate the role of high-dose araC in induction, of G-CSF priming, and of autologous stem cell transplantation.

DETAILED DESCRIPTION:
The present study by the German AML Cooperative Group has been designed in order to investigate the effects of AML typical therapeutic strategies for AML and related diseases. Thus, the entry criteria are age starting from 16 years with no upper age limit, de novo AML or AML secondary to chemotherapy or radiotherapy of another disease or myelodysplasia subtype RAEB with bone marrow blasts greater than 10 %. All randomization is stratified according to karyotype favorable / intermediate / unfavorable. Additional stratification is according to LDH </>= 700 U and age </>= 60 Y. Standard treatment is (A) double induction with TAD and HAM, consolidation with TAD and maintenance treatment with monthly AD-AT-AC-AT -, rotatingly. Experimental modifications to be compared with stan-dard treatment are (B) double induction with HAM-HAM, (C) multiple course G-CSF before and during chemotherapy courses and (D) instead of maintenance treatment myeloablative consolidation with Bu/Cy and autologous blood stem cell transplantation. Intent to treat conditions are guaranteed by randomization before induction treatment starts. In order to evaluate the effect of every single modification randomization to (C) is equally distributed to the patients in treatment arms (A) and (B) which is also true for the randomization to (D) (balanced randomization). Similarly balanced between treatment arms are the patients according to diagnosis, age and risk factors like serum LDH and karyotype. In order to adapt treatment intensity to age patients of 60 years and older receive the second induction course only in case of 5 % or more residual bone marrow blasts. In addition, the AraC dose in HAM is reduced to 1 instead of 3 g/sqm in this age group. Furthermore, there is no treatment arm including stem cell transplantation in patients of 60+ years. Pri-mary endpoint to compare the therapeutic strategies is event-free survival from treatment start (A, B, C) and from achievement of remission (D), respectively.

By this design the AMLCG 2000 trial can contribute relevant experiences on optimum therapeutic strategies for the biological subgroups of de novo AML, secondary AML and MDS. Furthermore, new biological subgroups and their significance related to treatment strategies can be defined.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (de-novo AML, secondary AML, high-risk MDS)
* Age 16 - no upper age limit
* Written informed consent

Exclusion Criteria:

* Severe comorbidity
* Presence of other malignancy
* Prior anti-leukemic treatment
* Pregnancy
* Severe psychiatric disorder or other circumstances which may compromise cooperation of the patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3500 (Actual)
Dates: Start 1999-06; Primary Completion 2007-01 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Remission rate, Remission duration,Relapse-free survival, Overall survival, Event-free survival | 12-18months

SECONDARY OUTCOMES:
Time and dose compliance, Realisation of SCT, Toxicity according to WHO | 12-18months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Buechner, MD PhD, Study Chair — University of Muenster, Medical Center, Department of Medicine, Hematology and Oncology
Locations (1):
- University of Muenster, Medical Center, Department of Medicine, Hematology and Oncology, Münster, Germany

REFERENCES:
- [Derived] Kunadt D, Stasik S, Metzeler KH, Rollig C, Schliemann C, Greif PA, Spiekermann K, Rothenberg-Thurley M, Krug U, Braess J, Kramer A, Hochhaus A, Scholl S, Hilgendorf I, Brummendorf TH, Jost E, Steffen B, Bug G, Einsele H, Gorlich D, Sauerland C, Schafer-Eckart K, Krause SW, Hanel M, Hanoun M, Kaufmann M, Wormann B, Kramer M, Sockel K, Egger-Heidrich K, Herold T, Ehninger G, Burchert A, Platzbecker U, Berdel WE, Muller-Tidow C, Hiddemann W, Serve H, Stelljes M, Baldus CD, Neubauer A, Schetelig J, Thiede C, Bornhauser M, Middeke JM, Stolzel F; A. M. L. Cooperative Group (AMLCG), Study Alliance Leukemia (SAL). Impact of IDH1 and IDH2 mutational subgroups in AML patients after allogeneic stem cell transplantation. J Hematol Oncol. 2022 Sep 5;15(1):126. doi: 10.1186/s13045-022-01339-8. PMID 36064577
- [Derived] Konstandin NP, Pastore F, Herold T, Dufour A, Rothenberg-Thurley M, Hinrichsen T, Ksienzyk B, Tschuri S, Schneider S, Hoster E, Berdel WE, Woermann BJ, Sauerland MC, Braess J, Bohlander SK, Klein HG, Hiddemann W, Metzeler KH, Spiekermann K. Genetic heterogeneity of cytogenetically normal AML with mutations of CEBPA. Blood Adv. 2018 Oct 23;2(20):2724-2731. doi: 10.1182/bloodadvances.2018016840. PMID 30337300
- [Derived] Prassek VV, Rothenberg-Thurley M, Sauerland MC, Herold T, Janke H, Ksienzyk B, Konstandin NP, Goerlich D, Krug U, Faldum A, Berdel WE, Wormann B, Braess J, Schneider S, Subklewe M, Bohlander SK, Hiddemann W, Spiekermann K, Metzeler KH. Genetics of acute myeloid leukemia in the elderly: mutation spectrum and clinical impact in intensively treated patients aged 75 years or older. Haematologica. 2018 Nov;103(11):1853-1861. doi: 10.3324/haematol.2018.191536. Epub 2018 Jun 14. PMID 29903761
- [Derived] Pastore F, Greif PA, Schneider S, Ksienzyk B, Mellert G, Zellmeier E, Braess J, Sauerland CM, Heinecke A, Krug U, Berdel WE, Buechner T, Woermann B, Hiddemann W, Spiekermann K. The NPM1 mutation type has no impact on survival in cytogenetically normal AML. PLoS One. 2014 Oct 9;9(10):e109759. doi: 10.1371/journal.pone.0109759. eCollection 2014. PMID 25299584
- [Derived] Herold T, Metzeler KH, Vosberg S, Hartmann L, Rollig C, Stolzel F, Schneider S, Hubmann M, Zellmeier E, Ksienzyk B, Jurinovic V, Pasalic Z, Kakadia PM, Dufour A, Graf A, Krebs S, Blum H, Sauerland MC, Buchner T, Berdel WE, Woermann BJ, Bornhauser M, Ehninger G, Mansmann U, Hiddemann W, Bohlander SK, Spiekermann K, Greif PA. Isolated trisomy 13 defines a homogeneous AML subgroup with high frequency of mutations in spliceosome genes and poor prognosis. Blood. 2014 Aug 21;124(8):1304-11. doi: 10.1182/blood-2013-12-540716. Epub 2014 Jun 12. PMID 24923295
- [Derived] Hubmann M, Kohnke T, Hoster E, Schneider S, Dufour A, Zellmeier E, Fiegl M, Braess J, Bohlander SK, Subklewe M, Sauerland MC, Berdel WE, Buchner T, Wormann B, Hiddemann W, Spiekermann K. Molecular response assessment by quantitative real-time polymerase chain reaction after induction therapy in NPM1-mutated patients identifies those at high risk of relapse. Haematologica. 2014 Aug;99(8):1317-25. doi: 10.3324/haematol.2014.104133. Epub 2014 May 9. PMID 24816240
- [Derived] Stelljes M, Krug U, Beelen DW, Braess J, Sauerland MC, Heinecke A, Ligges S, Sauer T, Tschanter P, Thoennissen GB, Berning B, Kolb HJ, Reichle A, Holler E, Schwerdtfeger R, Arnold R, Scheid C, Muller-Tidow C, Woermann BJ, Hiddemann W, Berdel WE, Buchner T. Allogeneic transplantation versus chemotherapy as postremission therapy for acute myeloid leukemia: a prospective matched pairs analysis. J Clin Oncol. 2014 Feb 1;32(4):288-96. doi: 10.1200/JCO.2013.50.5768. Epub 2013 Dec 23. PMID 24366930
- [Derived] Opatz S, Polzer H, Herold T, Konstandin NP, Ksienzyk B, Zellmeier E, Vosberg S, Graf A, Krebs S, Blum H, Hopfner KP, Kakadia PM, Schneider S, Dufour A, Braess J, Sauerland MC, Berdel WE, Buchner T, Woermann BJ, Hiddemann W, Spiekermann K, Bohlander SK, Greif PA. Exome sequencing identifies recurring FLT3 N676K mutations in core-binding factor leukemia. Blood. 2013 Sep 5;122(10):1761-9. doi: 10.1182/blood-2013-01-476473. Epub 2013 Jul 22. PMID 23878140
- [Derived] Buchner T, Schlenk RF, Schaich M, Dohner K, Krahl R, Krauter J, Heil G, Krug U, Sauerland MC, Heinecke A, Spath D, Kramer M, Scholl S, Berdel WE, Hiddemann W, Hoelzer D, Hehlmann R, Hasford J, Hoffmann VS, Dohner H, Ehninger G, Ganser A, Niederwieser DW, Pfirrmann M. Acute Myeloid Leukemia (AML): different treatment strategies versus a common standard arm--combined prospective analysis by the German AML Intergroup. J Clin Oncol. 2012 Oct 10;30(29):3604-10. doi: 10.1200/JCO.2012.42.2907. Epub 2012 Sep 10. PMID 22965967
- [Derived] Greif PA, Dufour A, Konstandin NP, Ksienzyk B, Zellmeier E, Tizazu B, Sturm J, Benthaus T, Herold T, Yaghmaie M, Dorge P, Hopfner KP, Hauser A, Graf A, Krebs S, Blum H, Kakadia PM, Schneider S, Hoster E, Schneider F, Stanulla M, Braess J, Sauerland MC, Berdel WE, Buchner T, Woermann BJ, Hiddemann W, Spiekermann K, Bohlander SK. GATA2 zinc finger 1 mutations associated with biallelic CEBPA mutations define a unique genetic entity of acute myeloid leukemia. Blood. 2012 Jul 12;120(2):395-403. doi: 10.1182/blood-2012-01-403220. Epub 2012 May 30. PMID 22649106
- [Derived] Stelljes M, Beelen DW, Braess J, Sauerland MC, Heinecke A, Berning B, Kolb HJ, Holler E, Schwerdtfeger R, Arnold R, Spiekermann K, Muller-Tidow C, Serve HL, Silling G, Hiddemann W, Berdel WE, Buchner T, Kienast J; German AML Cooperative Group (AMLCG). Allogeneic transplantation as post-remission therapy for cytogenetically high-risk acute myeloid leukemia: landmark analysis from a single prospective multicenter trial. Haematologica. 2011 Jul;96(7):972-9. doi: 10.3324/haematol.2011.041004. Epub 2011 Apr 1. PMID 21459795
- [Derived] Lin YH, Kakadia PM, Chen Y, Li YQ, Deshpande AJ, Buske C, Zhang KL, Zhang Y, Xu GL, Bohlander SK. Global reduction of the epigenetic H3K79 methylation mark and increased chromosomal instability in CALM-AF10-positive leukemias. Blood. 2009 Jul 16;114(3):651-8. doi: 10.1182/blood-2009-03-209395. Epub 2009 May 14. PMID 19443658